CLINICAL TRIAL: NCT04809584
Title: 18F-DCFPyL PET/MRI for Detection of Regional Nodal and Distant Metastases in Patients With Intermediate and High-risk Prostate Cancer
Brief Title: 18F-DCFPyL PET/MRI in Regional Nodal&Distant Metastases Detection in Intermediate &HR Prostate Cancer
Status: Approved for marketing | Type: Expanded Access
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-58503; PROS0103 (Other: OnCore); IRB-58503 (Other: Stanford IRB)
Record Dates: First submitted 2021-03-15; First posted 2021-03-22 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid; Gadolinium; motexafin gadolinium; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: F18-DCFPyL — Participant will be injected iv with 9 mCi ± 20% of 18F-DCFPyL
Drug: Gadolinium — Contrast agent
  Other Names: motexafin gadolinium
Procedure: Positron emission tomography (PET)/Magnetic Resonance Imaging (MRI) Scan — Imaging test that combines PET (positron emission tomography) and MRI (magnetic resonance imaging)

SUMMARY:
The purpose of this research study is to see if patients' tumor can be identified by 18F-DCFPyL PET/MRI scan. The radioactive study agent, 18FDCFPyL, combined with PET/MRI scan may be able to identify smaller tumors than the standard of care contrast-enhanced CT or MRI scan.

DETAILED DESCRIPTION:
This is an expanded access study with a total of 100 participants with newly diagnosed intermediate or high-risk prostate cancer scheduled to undergo prostatectomy and lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is older than 18-year-old
2. Biopsy proven prostate adenocarcinoma
3. Planned prostatectomy with lymph node dissection
4. Intermediate to high-risk disease (as determined by elevated Prostate-specific antigen (PSA) [PSA>10], T-stage [T2b or greater], Gleason score [Gleason score > 6] or other risk factors)
5. Able to provide written consent
6. Karnofsky performance status of ³50 (or Eastern Cooperative Oncology Group (ECOG) /World Health Organization (WHO) equivalent)

Exclusion Criteria:

1. Neoadjuvant chemotherapy or radiation therapy prior to prostatectomy including focal ablation techniques (HiFu)
2. Androgen deprivation therapy or other neoadjuvant treatments prior to PET imaging surgery
3. Metallic implants (contraindicated for MRI)

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Men >/= 18 years of age will be recruited.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei H Iagaru, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States